CLINICAL TRIAL: NCT00555997
Title: A 12-Week, Randomized, Double-Blind, Placebo-Controlled, Parallel-Sequential Trial of Ziprasidone as Monotherapy for Major Depressive Disorder
Brief Title: A 12-Week, Placebo Controlled Trial of Ziprasidone as Monotherapy for Major Depressive Disorder
Acronym: Geodon
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Cambridge Health Alliance (Other); University of Connecticut (Other); Vanderbilt University (Other); Psychiatric Medicine Associates, L.L.C. (Other); Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, George I. Papakostas, Director of Treatment-Resistant Studies, Depression Clinical and Research Program, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2007-P-000623; NCT00657592 (obsolete NCT alias)
Record Dates: First submitted 2007-11-07; First posted 2007-11-09 (Estimated); Results first posted 2014-07-03 (Estimated); Last update posted 2014-07-03 (Estimated); Status verified 2014-06

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Major Depression; Depression; Geodon; Ziprasidone
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — ziprasidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Patients in group 1 will receive Ziprasidone for the full 12 weeks of the study.
  Interventions: Drug: Ziprasidone
- 2 (Active Comparator): Patients in Group 2 will receive placebo for the first 6 weeks of the study, then will receive Ziprasidone for the last 6 weeks.
  Interventions: Drug: Ziprasidone
- 3 (Placebo Comparator): Patients in Group 3 will receive placebo for the full 12 weeks of the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ziprasidone — 20mg-80mg a day. Dose increases of 20mg per day may occur at three study visits as directed by clinician. Maximum; 80mg per day per patient.
  Other Names: Geodon
  Arms: 1
Drug: Ziprasidone — 20mg-80mg a day. Dose increases of 20mg per day may occur at three study visits as directed by clinician. Maximum; 80mg per day per patient.
  Other Names: Geodon
  Arms: 2
Drug: Placebo — 0mg Placebo per day. "Dose increases" and "dose decreases" may occur, but patient will remain at 0mg placebo
  Arms: 3

SUMMARY:
This is a study on the effectiveness, tolerability and safety of oral ziprasidone as monotherapy in patients with major depressive disorder (MDD). Outpatients suffering from MDD will be treated with either ziprasidone or placebo for 12 weeks.

Hypothesis: There will be a statistically significant difference in the magnitude of response, as measured by a decrease in baseline 17-item Hamilton Depression Rating Scale (HAM-D-17) scores, between the two treatment groups; the reduction in HAM-D-17 scores will be greater in the ziprasidone monotherapy group than in the placebo group.

DETAILED DESCRIPTION:
Exploratory hypothesis 1: There will be a statistically significant difference in the percentage of responders in the two treatment groups; response rates will be significantly higher for the ziprasidone monotherapy compared to the placebo group.

Exploratory hypothesis 2: The change in 6-VAS-D scores during the trial will be highly correlated to the change in HAM-D-17 and QIDS-SR during the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65.
2. Written informed consent.
3. MDD, current according to the fourth version of the Diagnostic and Statistical Manual for Mental Disorders (DSM-IV) as diagnosed by the Mini International Neuropsychiatric Interview (MINI; Sheehan et al, 1998).
4. Quick Inventory of Depressive Symptomatology - Self-Rated (QIDS-SR- Trivedi et al, 2004) score of at least 10 at both screen and baseline visits.

Exclusion Criteria:

1. Pregnant women.
2. Women of child bearing potential who are not using a medically accepted means of contraception (to include oral contraceptive or implant, condom, diaphragm, spermicide, intrauterine device, tubal ligation, or a partner with vasectomy).
3. Treatment with antidepressants for 2 weeks prior to the screen visit. If interested in discontinuing their current medication, potential participants must discuss this possibility with the prescribing physician. Study doctors will not implement any form of treatment washout.
4. Patients who no longer meet DSM-IV criteria for MDD during the baseline visit, or patients who demonstrate a 25% or greater reduction in QIDS-SR scores, screening to baseline.
5. Serious suicide or homicide risk, as assessed by the evaluating clinician or a score of 4 on the third item of the HAM-D.
6. Unstable medical illness including cardiovascular, hepatic, renal, respiratory, endocrine, neurological, or hematological disease.
7. Patients who meet criteria for alcohol or substance dependence, active within the last month.
8. Any bipolar disorder (current or past).
9. Any psychotic disorder (current or past).
10. Psychotic features in the current episode or a history of psychotic features.
11. History of a seizure disorder.
12. Clinical or laboratory evidence of untreated hypothyroidism.
13. Patients requiring excluded medications (see table 1 for details).
14. Prior course of ziprasidone, or intolerance to ziprasidone at any dose.
15. Any investigational psychotropic drug within the last 3 months.
16. Patients with significant cardiac conduction problems on screening electrocardiogram such as atrial fibrillation, atrial flutter, atrio-ventricular block, prolonged or abnormal QTc interval (i.e. QTc>450msec), or prolonged QRS interval.
17. Patients who have suffered a myocardial infarction within the past 12 months, with uncompensated heart failure, or a history of QTc prolongation.
18. Patients with abnormal serum potassium or magnesium levels upon screening.
19. Patients currently taking other drugs that prolong the QTc including dofetilide, sotalol, quinidine, class Ia antiarrhythmics, class III antiarrhythmics, mesoridazine, thioridazine, chlorpromazine, droperidol, pimozide, sparfloxacin, gatifloxacin, moxifloxacin, halofantrine, mefloquine, pentamidine, arsenic trioxide, levomethadyl acetate, dolasetron methylate, probucol or tacrolimus.
20. Patients who have failed to experience significant clinical improvement following 3 or more antidepressant trials of adequate duration (at least 6 weeks) and dose (minimal effective doses defined as: fluoxetine, paroxetine, citalopram 20mg; sertraline, fluvoxamine 50mg, escitalopram 10mg, paroxetine CR 25mg, venlafaxine 75mg, duloxetine 60mg, bupropion 150mg, 15mg of mirtazapine, trazodone or nefazodone 300mg).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George I Papakostas, M.D., Principal Investigator — Massachusetts General Hospital; John M Zajecka, M.D., Principal Investigator — Psychiatric Medicine Associates, L.L.C.; Richard C Shelton, M.D., Principal Investigator — Vanderbilt University Medical Center; Andrew Winokur, M.D., Principal Investigator — UConn Health; Gustavo Kinrys, M.D., Principal Investigator — Cambridge Health Alliance; Waguih IsHak, M.D., Principal Investigator — Cedar's Sinai; Mahmoud S Okasha, MD, Principal Investigator — Comprehensive Psychiatric Care, Norwich CT
Locations (7):
- United States (7):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Connecticut Health Center, Farmington, Connecticut
  - Comprehensive Psychiatric Care, Norwich, Connecticut
  - Psychiatric Medicine Associates, L.L.C., Chicago, Illinois
  - Massachusetts General Hosptial, Boston, Massachusetts
  - Cambridge Health Alliance, Cambridge, Massachusetts
  - Vanderbilt University Medical Center, Nashville, Tennessee

REFERENCES:
- [Result] Papakostas GI, Vitolo OV, Ishak WW, Rapaport MH, Zajecka JM, Kinrys G, Mischoulon D, Lipkin SH, Hails KA, Abrams J, Ward SG, Meisner A, Schoenfeld DA, Shelton RC, Winokur A, Okasha MS, Bari MA, Fava M. A 12-week, randomized, double-blind, placebo-controlled, sequential parallel comparison trial of ziprasidone as monotherapy for major depressive disorder. J Clin Psychiatry. 2012 Dec;73(12):1541-7. doi: 10.4088/JCP.12m07670. PMID 23290327
- [Derived] Heo JY, Jeon HJ, Fava M, Mischoulon D, Baer L, Clain A, Doorley J, Pisoni A, Papakostas GI. Efficacy of ziprasidone monotherapy in patients with anxious depression: a 12-week, randomized, double-blind, placebo-controlled, sequential-parallel comparison trial. J Psychiatr Res. 2015 Mar;62:56-61. doi: 10.1016/j.jpsychires.2015.01.007. Epub 2015 Jan 26. PMID 25659187

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1 Ziprasidone: Subjects taking ziprasidone in the first phase.
- Phase 1 Placebo: Subjects taking placebo in the first phase.
- Phase 2 Ziprasidone: Subjects taking ziprasidone in the second phase.
- Phase 2 Placebo: Patients who received placebo in phase 2.
Period: Phase 1 SPCD
Arm/Group | Phase 1 Ziprasidone | Phase 1 Placebo | Phase 2 Ziprasidone | Phase 2 Placebo
Started | 29 | 91 | 0 | 0
Completed | 17 | 76 | 0 | 0
Not Completed | 12 | 15 | 0 | 0
Period: Phase 2 SPCD
Arm/Group | Phase 1 Ziprasidone | Phase 1 Placebo | Phase 2 Ziprasidone | Phase 2 Placebo
Started | 0 | 0 | 38 | 25
Completed | 0 | 0 | 31 | 22
Not Completed | 0 | 0 | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Placebo/Ziprasidone: Received placebo in first phase and ziprasidone in second phase
- Placebo: Subjects received placebo throughout study
- Ziprasidone: Subjects received ziprasidone throughout study
- Total: Total of all reporting groups
Arm/Group | Placebo/Ziprasidone | Placebo | Ziprasidone | Total
Number analyzed (Participants) | 47 | 44 | 29 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 47 | 42 | 29 | 118
  >=65 years | 0 | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.1 (11.1) | 44.6 (11.0) | 41.5 (10.6) | 43.7 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 22 | 13 | 53
  Male | 29 | 22 | 16 | 67
Region of Enrollment [Number; unit: participants]
  United States | 47 | 44 | 29 | 120

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Rating Scale (HAM-D-17) Scores
Description: Higher numbers represent more symptoms of a major depressive episode. Minimum is 0. Maximum is 52.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: points
Groups:
- Ziprasidone Phase I: Results from phase I for those taking ziprasidone during that phase
- Placebo Phase I: Results from phase I for those taking placebo during that phase
- Ziprasidone Phase II: Results from phase II for those taking ziprasidone during that phase
- Placebo Phase II: Results from phase II for those taking placebo during that phase
Arm/Group | Ziprasidone Phase I | Placebo Phase I | Ziprasidone Phase II | Placebo Phase II
Number analyzed (Participants) | 29 | 91 | 21 | 25
points
  Mean phase baseline score | 20.1 (5.5) | 19.9 (4.8) | 14.7 (3.9) | 15.6 (5.9)
  Mean phase score reduction | -8.8 (7.3) | -7.1 (7.0) | -2.1 (5.2) | -4.3 (6.0)

2. Secondary Outcome: Responder/Non-responder
Description: A responder during phase 1 or phase 2 is someone who demonstrated a 50% or greater decrease in HAMD-17 scores during phase 1 or phase 2 (corresponding).
Time Frame: 6 weeks
Measure: Number; unit: percentage of patients
Arm/Group | Ziprasidone Phase I | Placebo Phase I | Ziprasidone Phase II | Placebo Phase II
Number analyzed (Participants) | 29 | 91 | 21 | 25
percentage of patients | 44.8 | 31.8 | 23.8 | 28.0

3. Secondary Outcome: Change in 6-VAS-D Scores During Each Phase.
Time Frame: 6 weeks
Population: Forms not analyzable due to insufficient standardization across sites.
Arm/Group | Phase 1 Ziprasidone | Phase 1 Placebo | Phase 2 Ziprasidone | Phase 2 Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year, 4 months
Groups:
- Ziprasidone: Adverse events experienced by subjects while taking ziprasidone
- Placebo: Adverse events experienced when taking placebo
Arm/Group | Ziprasidone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/80 | 1/125
Other Adverse Events (participants affected / at risk) | 31/125 | 22/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ziprasidone (N=80) | Placebo (N=125)
Hospitalization due to suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ziprasidone (N=125) | Placebo (N=80)
Sedation/Fatigue (Psychiatric disorders) | 13 | 3
Headache (Nervous system disorders) | 3 | 2
Insomnia (Psychiatric disorders) | 2 | 3
Dizziness (Nervous system disorders) | 2 | 2
Blurry/Double Vision (Nervous system disorders) | 2 | 2
Akathisia/Agitation (Psychiatric disorders) | 1 | 1
Dry mouth (Gastrointestinal disorders) | 6 | 6
Constipation (Gastrointestinal disorders) | 3 | 3
Increased appetite (Gastrointestinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 1 | 2
Weight gain (Gastrointestinal disorders) | 0 | 1
Sexual dysfunction (General disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No